CLINICAL TRIAL: NCT00855062
Title: Minocycline in the Treatment of HIV-Associated Cognitive Impairment in Uganda
Brief Title: Minocycline for HIV+ Cognitive Impairment in Uganda
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Neurologic AIDS Research Consortium Data Safety and Monitoring Board committee recommended to terminate the study early due to futility on 11/6/2009.
Sponsor: Johns Hopkins University (Other)
Collaborators: Makerere University (Other)
Responsible Party: Ned Sacktor, MD, Johns Hopkins School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uganda minocycline study; Grant Number: 5 UO1 NS32228
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-01

CONDITIONS: HIV-associated Cognitive Impairment; HIV Infections
Keywords: Human immunodeficiency virus (HIV); HIV associated cognitive impairment; HIV dementia; Uganda; Acquired immune deficiency syndrome (AIDS); Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS Dementia Complex | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Active Comparator): Minocycline 100 mg orally every 12 hours
  Interventions: Drug: minocycline
- Placebo (Placebo Comparator): Placebo minocycline capsules every 12 hours
  Interventions: Drug: minocycline placebo capsule

INTERVENTIONS:
Drug: minocycline — 100 mg capsule every 12 hours by mouth
  Arms: Minocycline
Drug: minocycline placebo capsule — 1 capsule every 12 hours by mouth
  Arms: Placebo

SUMMARY:
Purpose: The purpose of the study is to assess the safety and effectiveness of minocycline, an antibiotic, in the treatment of Human immunodeficiency virus (HIV)-associated cognitive impairment in Uganda.

Study Design: Treatment, 24-week Randomized, Placebo-Controlled, Double-Blind Phase with Optional 24-week Open Label Phase for Subjects with a cluster of differentiation 4 (CD4) Count in the 251-350 Range

* Arm 1: Minocycline 100 mg orally every 12 hours (50 subjects)
* Arm 2: Matching placebo orally every 12 hours (50 subjects)

Primary Objective:

· To examine whether minocycline treatment will improve cognitive performance after 24 weeks compared to baseline

Secondary Objectives:

* To examine whether minocycline treatment for 24 weeks is safe and well-tolerated in individuals with HIV-associated cognitive impairment
* To examine whether minocycline treatment for 48 weeks is safe and well-tolerated in individuals with HIV-associated cognitive impairment
* To examine whether minocycline treatment for 24 weeks improves functional impairment

ELIGIBILITY:
Inclusion Criteria:

* HIV infection prior to study entry
* Naïve to any antiretroviral regimen and ineligible to receive antiretroviral therapy by cluster of differentiation 4 (CD4) criteria in Uganda
* Negative serum or urine pregnancy test for women of childbearing potential
* Willingness to use birth control
* Age 18-65 years
* AIDS Dementia Scale Stage 0.5 OR 1
* Impaired cognitive performance as evidenced by an International HIV Dementia Scale (HDS) as defined by the protocol
* Ability to sit or stand and swallow intact capsules with an 8-ounce glass of water
* Ability and willingness of subject or legal guardian/ representative to give written informed consent
* Resident within a 20km radius of Kampala city

Exclusion Criteria:

* Current cancers other than basal cell carcinoma, in situ carcinoma of the cervix, or Kaposi's sarcoma without evidence of visceral involvement or which does not require systemic chemotherapy
* Severe premorbid psychiatric illness, including schizophrenia and major depression which, in the in investigator's opinion, is likely to interfere with study compliance
* Active symptomatic AIDS-defining opportunistic infection within 45 days prior to study entry
* Confounding neurological disorders as defined in the protocol
* Central nervous system infections or cancers as defined in the protocol
* Systemic lupus
* Thyroid disease diagnosed within 24 weeks prior to entry
* Breastfeeding
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator
* History of allergy/sensitivity to minocycline or other tetracyclines and their formulations
* Any other clinically significant condition or laboratory abnormality that, in the opinion of the investigator, would interfere with the subject's ability to participate in the study. This includes an individual found to have an HIV dementia scale stage 3 or 4.
* Any esophageal or other condition that would interfere with the swallowing of the study medication
* Use of excluded drugs as defined by the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ned Sacktor, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Infecious Diseas Institute, Kampala, Uganda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from Mar 2008 to Oct 2009 when the study was stopped early (Data and Safety Monitoring Board (DSMB) decision based on futility) on Nov 2009. The study participants were recruited from the Infectious Disease Institute, Makerere University, Kampala, Uganda.
Pre-assignment Details: Total of 353 participants were screened; only 73 were randomized and thus 280 were not enrolled: 146 of them did not have cognitive impairment, 55 of them lacked laboratory inclusion criteria, and 79 of them had "others".
Period: Step1
Arm/Group | Minocycline | Placebo
Started | 36 | 37
Completed | 26 | 26
Not Completed | 10 | 11
Not completed — Early Study Closure | 5 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Period: Step2
Arm/Group | Minocycline | Placebo
Started | 19 (26 participants completed STEP1; however, only 19 out of the 26 decided to enroll in STEP2.) | 21 (26 participants completed STEP1; however, only 21 out of the 26 decided to enroll in STEP2.)
Completed | 13 | 15
Not Completed | 6 | 6
Not completed — Early Study Closure | 6 | 2
Not completed — Adverse Event | 0 | 3
Not completed — Initiation of antiretroviral therapy/ART | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 37 | 73
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (8.21) | 36.7 (7.17) | 37.0 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Uganda | 36 | 37 | 73
Baseline Memorial Sloan Kettering (MSK) Acquired Immune Deficiency Syndrome (AIDS) Dementia Scale [Number; unit: Participants] — The Memorial Sloan Kettering (MSK) clinical scale was defined below:
  * Stage 0: normal
  * Stage 0.5: equivocal/subclinical
  * Stage 1: mild
  * Stage 2: moderate
  * Stage 3: severe
  * Stage 4: end stage
  Participants
    Equivocal/subclinical | 35 | 37 | 72
    Mild | 1 | 0 | 1
Baseline Cluster of Differentiation Four (CD4) Count [Median (Full Range); unit: cells/mm^3] | 319 [251 to 469] | 305 [252 to 500] | 313 [251 to 500]
Baseline Log10(Human immunodeficiency virus (HIV) Ribonucleic Acid (RNA) Viral Load (VL)) [Log Mean (Inter-Quartile Range); unit: copies/mL] | 4.41 [4.09 to 4.94] | 4.59 [4.12 to 5.25] | 4.50 [4.10 to 5.10]
Baseline Karnofsky's Performance Score [Number; unit: Participants] — 100:Normal,90:normal;Minor Signs or Symptoms of Disease,80:Normal Activity with Effort;Some Signs or Symptoms of Disease,70:Cares for Self,Unable to Carry on Normal Activity or to Do Active Work,60:Requires Occasional Assistance but is Able to Care for Most of Needs,50:Requires Considerable Assistance and Frequent Medical Care,40:Disabled,Requires Special Care and Assistance,30:Severely Disabled; Hospitalization Indicated Although Death is Not Imminent,20:Very Sick; Hospitalization Necessary;Active Supportive Treatment is Necessary,10:Moribund, Fatal Processes Progressing Rapidly,0:Death
  Participants
    80 (Karnofsky Score) | 1 | 2 | 3
    90 (Karnofsky Score) | 35 | 34 | 69
    100 (Karnofsky Score) | 0 | 1 | 1
Baseline Instrumental Activities of Daily Living (IADL) [Number; unit: Participants] — 16 tasks: Housekeeping,Managing Finances,Buying Groceries,Cooking,Planning Social Activities,Understanding Reading Materials/TV,Transportation,Using the Telephone,Home Repairs,Bathing,Dressing,Shopping,Laundry,Taking/Keeping Track of Medication,Child Care,Work.
  For the baseline IADL measure, participants were given four choices to choose for having difficulty on the 16 tasks:Primarily Cognitive problems,Primarily physical problems,equally cognitive and physical problems,not having any difficulties on previous tasks.
  Participants
    Primarily cognitive problems | 1 | 0 | 1
    Primarily physical problems | 6 | 2 | 8
    Not having any difficulties on the tasks | 29 | 35 | 64
Baseline Overall Neurological Assessment [Number; unit: Participants]
  Normal neurological assessment | 26 | 30 | 56
  Central Nervous System (CNS) abnormality only | 4 | 5 | 9
  Peripheral Nervous System (PNS) abnormality only | 4 | 1 | 5
  CNS and PNS abnormality | 1 | 1 | 2
  Can not assess | 1 | 0 | 1
Baseline Uganda Neuropsychological Test Battery Summary measure (U NP Sum) [Mean (Standard Deviation); unit: z-scores] — Uganda Neuropsychological Test Battery Summary measure (U NP Sum)is the average z-scores of the 9 neurupsychological tests:Grooved Pegboard Dominant Hand,Grooved Pegboard Non-dominant Hand,Color Trail1,Color Trail2,Symbol Digit,WHO/UCLA Verbal Learning Test Trial 5,WHO/UCLA Verbal Learning Test Delayed Recall,Digit Span-Forward,Digit Span-Backward Since the score depends on age and education levels, the raw score was standardized as follows: Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -0.97 (0.78) [-1.16 to -0.55] | -0.97 (0.86) [-1.18 to -0.58] | -0.97 (0.82) [-1.18 to -0.55]
WHO-UCLA Auditory Verbal Learning Test (AVLT): Trials Total [Mean (Standard Deviation); unit: z-scores] — World Health Organization-University of California Los Angeles (WHO-UCLA) Auditory Verbal Learning Test (AVLT) is a full-scale memory assessment.
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -1.28 (0.88) | -1.48 (1.14) | -1.38 (1.02)
WHO-UCLA Auditory Verbal Learning Test (AVLT): Delayed [Mean (Standard Deviation); unit: z-scores] — World Health Organization-University of California Los Angeles (WHO-UCLA) Auditory Verbal Learning Test (AVLT) is a memory assessment.
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -1.17 (0.79) | -1.15 (1.18) | -1.16 (1.00)
Color Trails 1 [Mean (Standard Deviation); unit: z-scores] — The Color Trails tests measure speed of attention, sequencing, mental flexibility, visual search, and motor function.
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -1.35 (2.03) | -1.65 (3.03) | -1.51 (2.60)
Color Trails 2 [Mean (Standard Deviation); unit: z-scores] — The Color Trails tests measure speed of attention, sequencing, mental flexibility, visual search, and motor function.
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -2.55 (2.07) | -2.33 (2.05) | -2.44 (2.05)
Grooved Pegboard Dominant [Mean (Standard Deviation); unit: z-scores] — The grooved pegboard is a manipulative dexterity test requiring rapid visual-motor coordination. The test is completed using the dominant hand (GPD) and then using the non-dominant hand (GPN). The score for each hand is the time in seconds that the participant takes to complete the entire board.
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -0.34 (1.58) | -0.03 (1.14) | -0.18 (1.37)
Grooved Pegboard Non-dominant [Mean (Standard Deviation); unit: z-scores] — The grooved pegboard is a manipulative dexterity test requiring rapid visual-motor coordination. The test is completed using the dominant hand (GPD) and then using the non-dominant hand (GPN). The score for each hand is the time in seconds that the participant takes to complete the entire board.
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -0.56 (1.82) | -0.48 (1.42) | -0.52 (1.61)
Symbol Digit [Mean (Standard Deviation); unit: z-scores] — This test assesses the participant's ability to maintain rapid visual-motor sequencing in a timed test. The score is the total number of correctly transcribed numbers in the time limit (90 seconds). Participants receive 1 point for each item filled in correctly. Maximum score is 110 points.
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -0.87 (0.96) | -0.86 (0.80) | -0.86 (0.88)
Digit Span Backward [Mean (Standard Deviation); unit: z-scores] — Digit span assesses attention, concentration, and mental control(e.g., Repeat the numbers 1-2-3 in reverse sequence).
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | -0.68 (0.75) | -0.94 (1.06) | -0.81 (0.93)
Digit Span Forward [Mean (Standard Deviation); unit: z-scores] — Digit span assesses attention, concentration, and mental control(e.g., Repeat the numbers 1-2-3 in reverse sequence).
  Since the score depends on age and education levels, the raw score was standardized as follows:
  Zx =(x - μx)/σx where Zx is the age and education adjusted z-score, x is the raw score, and μx and σx are the age and education stratified norms.
  z-scores | 0.02 (0.79) | 0.19 (0.99) | 0.11 (0.90)

OUTCOME MEASURES:

1. Primary Outcome: 24-week Change of Uganda Neuropsychological Test Battery Summary Measure (U NP Sum)
Description: The U NP Sum is defined as the average of z scores for 9 neuropsychological test subcomponents in the neuropsychological test battery (i.e. the average of norm-adjusted ("z") scores for Grooved Pegboard Dominant Hand, Grooved Pegboard Non-dominant Hand, Color Trails 1, Color Trails 2, Symbol Digit, WHO-UCLA Verbal Learning test Trial 5, WHO-UCLA Verbal Learning test delayed recall, Digit Span forward and Digit Span backward). The outcome is defined as U NP Sum at week 24 - U NP Sum at baseline.
Time Frame: At baseline and week 24
Population: The descriptive statistics are based on per protocol analysis. For the statistical analysis, ITT analysis was used and the missing U NP Sums at week 24 were imputed using a multiple regression imputation method. The number of participants analyzed for the ITT analysis was 73 (36 for Minocycline and 37 for Placebo).
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 30 | 29
z-score | 0.44 (0.74) | 0.49 (0.67)
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis was that the 24-week changes of U NP Sum between the minocycline and placebo groups are the same. The sample size calculation showed that 100 (50 participants in each group) were required to detect the clinically meaningful difference of 0.5 with 85% power, 0.05 Type I error, two-sample and two-sided test; Test type: Superiority or Other; p = 0.370, Regression, Linear — The p-value was not adjusted for multiple comparisons; Slope = -0.026, 95% CI 2-sided [-0.512 to 0.460], Standard Error of Mean 0.248

2. Secondary Outcome: 24-week Change of Memorial Sloan Kettering (MSK) HIV Dementia Stage
Description: The outcome is a new dichotomous variable: no change/worse vs. better at 24 weeks compared to baseline.
Time Frame: At baseline and week 24
Population: The descriptive statistics were based on observed data. Since all participants reported there were no change in the MSK score at week 24, no statistical test was conducted.
Measure: Number; unit: participants
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 28 | 27
participants
  No Change/Worse | 28 | 27
  Better | 0 | 0

3. Secondary Outcome: 24-week Change of Karnofsky Performance Score
Description: The outcome is a new dichotomous variable: no change/worse vs. better at 24 weeks compared to baseline.
Time Frame: At baseline and week 24
Population: This analysis includes the participants with Karnofsky performance score at baseline and week 24.
Measure: Number; unit: percentage of participants
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 32 | 31
percentage of participants
  No Change/Worse | 97 | 94
  Better | 3 | 6
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the percentage of participants feeling "better" in the minocycline group after 24 week treatment is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.613, Fisher Exact — The p-value is not adjusted for multiple comparisons; Median Difference (Net) = 0.053, 95% CI 2-sided [0.043 to 0.062]

4. Secondary Outcome: Time From Treatment Initiation to the Development of a Grade ≥ 2 Toxicity and/or Sign and Symptoms.
Description: The outcome is the time to first Grade ≥ 2 toxicity and/or sign and symptoms from study treatment initiation up to week 24. The grade was determined by clinicians and an Grade ≥ 2 event means moderate, severe, life-threatening, or death event.
Time Frame: Time of initial Grade ≥ 2 toxicity and/or sign and symptom event up to week 24
Population: This analysis includes every randomized participants. A total of 21 minocycline and 20 placebo participants reported at least one Grade ≥ 2 toxicity and/or sign and symptoms during 24 weeks
Measure: Number; unit: participants with an event
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 36 | 37
participants with an event
  0-4 weeks | 12 | 10
  4.01 - 12 weeks | 6 | 7
  12.01 - 24 weeks | 3 | 3
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the survival curve for the first Grade ≥ 2 toxicity and/or sign and symptoms in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.661, Log Rank — The p-value is not adjusted for multiple comparisons

5. Secondary Outcome: Time From Treatment Initiation to the Development of a Grade ≥ 2 Toxicity and/or Sign and Symptoms
Description: The outcome is the time of first Grade ≥ 2 toxicity and/or sign and symptoms from treatment initiation up to 48 weeks. The grade was determined by clinicians and an Grade ≥ 2 event means moderate, severe, life-threatening, or death event.
Time Frame: Time of first Grade ≥ 2 toxicity and/or sign and symptom event up to 48 weeks
Population: This analysis includes every randomized participants. A total of 22 minocycline and 21 placebo participants reported at least one Grade ≥ 2 toxicity and/or sign and symptoms during 48 weeks.
Measure: Number; unit: participants with an event
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 36 | 37
participants with an event
  0-4 weeks | 12 | 10
  4.01-12 weeks | 6 | 7
  12.01-24 weeks | 3 | 3
  24.01-48 weeks | 1 | 1
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the 48-week survival curve for the first Grade ≥ 2 toxicity and/or sign and symptoms in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.941, Log Rank — The p-value is not adjusted for multiple comparisons

6. Secondary Outcome: 24-week Change of CD4 Cell Counts
Description: The outcome is defined as CD4 cell count at week 24 - CD4 cell count at baseline. The unit is cells/mm^3.
Time Frame: At baseline and week 24
Population: This analysis used the participants with CD4 cell counts at baseline and week 24.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 29 | 28
cells/mm^3 | -25.28 (70.85) | -28.57 (61.65)
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the mean 24-week change of CD4 cell counts in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.647, Regression, Linear — The p-value is not adjusted for multiple comparisons; The model was adjusted for the baseline CD4 counts; Mean Difference (Net) = 8.11, 95% CI 2-sided [-27.23 to 43.45], Standard Error of Mean 17.63

7. Secondary Outcome: 48-week Change of CD4 Cell Counts
Description: The outcome is defined as CD4 cell count at week 48 - CD4 cell count at baseline. The unit is cells/mm^3.
Time Frame: At baseline and week 48
Population: This analysis used the participants with CD4 cell counts at baseline and week 48.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 13 | 16
cells/mm^3 | -61.15 (80.46) | -56.50 (84.97)
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the mean 48-week change in CD4 cell counts in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.813, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the baseline CD4 counts; Mean Difference (Net) = 7.77, 95% CI 2-sided [-59.07 to 74.60], Standard Error of Mean 32.51

8. Secondary Outcome: 24-week Change of Instrumental Activities of Daily Living
Description: The outcome is a new dichotomous variable: no change/worse vs. better at 24 weeks compared to baseline.
Time Frame: At baseline and week 24
Population: The analysis includes participants with IADL scores at baseline and week 24.
Measure: Number; unit: percentage of participants
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 28 | 26
percentage of participants
  No Change/Worse | 86 | 88
  Better | 14 | 12
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the percentage of being "better" at week 24 compared to baseline in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.764, Regression, Logistic — The p-value is not adjusted for multiple comparisons; The model was not adjusted for any covariate (due to small number of being "better" in both groups; Odds Ratio (OR) = 1.28, 95% CI [0.26 to 6.34], Standard Error of Mean 0.82

9. Secondary Outcome: 24-week Change of HIV RNA Plasma Viral Loads (Log10 Transformed)
Description: The outcome is the HIV RNA plasma viral loads (Log10 transformed) at week 24 - the viral loads (Log10 transformed) at baseline.
Time Frame: At baseline and week 24
Population: The analysis includes participants with HIV RNA viral loads at baseline and week 24.
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 22 | 25
copies/mL | 0.22 [-0.14 to 0.50] | 0.13 [-0.23 to 0.43]
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the median log10-transformed HIV RNA viral loads in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.766, Kruskal-Wallis — The p-value is not adjusted for multiple comparisons; The chi-square score was 0.024 and the degree of freedom was 1

10. Secondary Outcome: 24-week Change of Center for Epidemiologic Studies Depression (CES-D) Score
Description: The outcome is the total CES-D score at week 24 - the total CES-D score at baseline.
  The total CES-D score is based on 20 CES-D items, such as "I was bothered by things that usually don't bother me" and "I did not feel like eating, my appetite was poor". Patients were asked to answer each item by 4 scales: (1) Rarely, (2) Sometimes, (3) Occasionally, and (4) Most of the time. After 4 negative items were multiplied by -1, the total CES-D score is a simple sum of all items.
  The min and Max are 0 and 60, respectively. Higher scores indicate more severe depressive symptoms.
Time Frame: At baseline and week 24
Population: The analysis includes participants with CES-D scores at baseline and week 24.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 31 | 28
scores on a scale | -4.19 (10.86) | -4.04 (8.27)
Statistical Analysis 1: Comparison: Minocycline vs Placebo; The null hypothesis is that the mean 24-week change of CES-D score in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.915, Regression, Linear — The p-value is not adjusted for multiple comparisons; The model was adjusted for the baseline CES-D and MSK scores; Mean Difference (Net) = 0.19, 95% CI 2-sided [-3.40 to 3.78], Standard Error of Mean 1.79

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: The lab assessments were conducted at weeks 0, 12, 24, and 48.
Arm/Group | Minocycline | Placebo
Serious Adverse Events (participants affected / at risk) | 2/36 | 1/37
Other Adverse Events (participants affected / at risk) | 26/36 | 25/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=36) | Placebo (N=37)
Death (Infections and infestations) | 1 (1) | 0 (0) — The patient died due to Pulmonary Tuberculosis. The cause of death was unrelated to the study treatment as she was not on the study treatment at the time of her death.
Potassium (Renal and urinary disorders) | 1 (1) | 0 (0) — The participant had high potassium level. The value was 7.8 when the normal limit was 5.3.
Sgpt (Hepatobiliary disorders) | 0 (0) | 1 (1) — The lab value was 836 when the normal value was 45.
Sgot (Hepatobiliary disorders) | 0 (0) | 1 (1) — The lab value was 901 when the normal value was 40.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=36) | Placebo (N=37)
Fever (General disorders) | 2 (2) | 1 (1)
Allergic Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Carbon Dioxide (General disorders) | 4 (4) | 2 (2)
Phosphorus (Renal and urinary disorders) | 3 (3) | 3 (3)
Sodium (Renal and urinary disorders) | 2 (2) | 1 (1)
Absolute Neutrophil Count (Blood and lymphatic system disorders) | 12 (21) | 12 (12)
SGOT (Hepatobiliary disorders) | 3 (3) | 0 (0)
White Blood Cells (Blood and lymphatic system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The estimated sample size was 100; however, due to early termination of the study, the total number of randomized participants was 73.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No